CLINICAL TRIAL: NCT00684307
Title: A Controlled, Randomized, Parallel, Multicentre Study to Assess Safety and Tolerability of the Oral Direct Thrombin Inhibitor AZD0837, Given as an Extended-release Formulation, in the Prevention of Stroke and Systemic Embolic Events in Patients With Atrial Fibrillation
Brief Title: Prevention of Stroke and Systemic Embolic Events in Patients With Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D1250C00008
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2011-09-22 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Nonvalvular Atrial Fibrillation
Keywords: Anticoagulant Treatment; Risk Factors For Stroke
MeSH Terms: interventions — AZD 0837; Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): AZD0837 450 mg
  Interventions: Drug: AZD0837
- 2 (Experimental): AZD0837 200 mg
  Interventions: Drug: AZD0837
- 3 (Experimental): AZD0837 300 mg
  Interventions: Drug: AZD0837
- 4 (Experimental): AZD0837 150 mg
  Interventions: Drug: AZD0837
- 5 (Active Comparator): Vitamin-K antagonist at INR 2-3
  Interventions: Drug: Vitamin-K antagonist at INR 2-3

INTERVENTIONS:
Drug: AZD0837 — ER tablet, PO, once daily for a period of 3-9 months.
  Arms: 1; 3; 4
Drug: Vitamin-K antagonist at INR 2-3 — Tablet, PO for a period of 3-9 months.
  Other Names: Warfarin
  Arms: 5
Drug: AZD0837 — ER tablet, PO, twice daily for a period of 3-9 months
  Arms: 2

SUMMARY:
The main purpose of this study is to provide dose-guiding information by assessing the safety and tolerability of 4 different dosing regimens of an extended-release (ER) formulation of AZD0837 compared with well-controlled, dose-adjusted Vitamin-K antagonists (VKA) (aiming for an international normalized ratio (INR) 2.0 to 3.0) in patients with non-valvular atrial fibrillation (AF) with one or more additional risk factors for stroke.

ELIGIBILITY:
Inclusion Criteria:

* Nonvalvular AF (NVAF) verified by at least two ECGs in the last year separated by at least one week.
* Previous cerebral ischemic attack (stroke or TIA, >30 days prior to randomization)
* Previous systemic embolism.
* Symptomatic congestive heart failure (CHF)
* Impaired left ventricular systolic function
* Diabetes mellitus
* Hypertension requiring anti-hypertensive treatment.

Exclusion Criteria:

* AF secondary to reversible disorders, eg hyperthyroidism, drugs and pulmonary embolism
* Known contraindication to VKA treatment
* Presence of a valvular heart disease, mechanical heart valves, active endocarditis, left ventricular aneurysm or thrombus, atrial myxoma or any condition other than AF requiring chronic anticoagulation treatment
* Conditions associated with increased risk of major bleeding for example: history of intracranial bleeding, history of bleeding gastrointestinal disorder or major surgical procedure or trauma two weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1084 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Y Lip, Prof, Principal Investigator — University Department of Medicine, City Hospital, Birmingham, B18 7QH, England, UK

REFERENCES:
- [Derived] Lip GY, Rasmussen LH, Olsson SB, Jensen EC, Persson AL, Eriksson U, Wahlander KF; Steering Committee. Oral direct thrombin inhibitor AZD0837 for the prevention of stroke and systemic embolism in patients with non-valvular atrial fibrillation: a randomized dose-guiding, safety, and tolerability study of four doses of AZD0837 vs. vitamin K antagonists. Eur Heart J. 2009 Dec;30(23):2897-907. doi: 10.1093/eurheartj/ehp318. Epub 2009 Aug 18. PMID 19690349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included male and female participants >18 years of age with chronic non-valvular Atrial Fibrillation. The participants were recruited during the time period from 20 February 2007 to 5 June 2008 at medical clinics in Europe.
Pre-assignment Details: Participants were enrolled in the study up to two weeks before randomisation and treatment assignment. Participants that were already treated with Vitamin K Antagonists (VKA) at the time of enrollment had their dose adjusted to achive INR <2.0 at the time of randomisation. If this was not achieved the participant was discontinued from the study.
Groups:
- 150 mg od: AZD0837 150 mg od
- 300 mg od: AZD0837 300 mg od
- 450 mg od: AZD0837 450 mg od
- 200 mg bd: AZD0837 200 mg bd
Period: Overall Study
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Started | 164 (Patients who received treatment) | 151 | 156 | 160 | 318
On Treatment Period Started | 164 | 151 | 156 | 160 | 318
On Treatment Period Completed | 140 (Patients who completed treatment) | 129 | 128 | 128 | 293
Completed | 140 | 129 | 128 | 128 | 293
Not Completed | 24 | 22 | 28 | 32 | 25
Not completed — Adverse Event | 11 | 6 | 15 | 16 | 8
Not completed — Development of increasing Liver Function | 0 | 2 | 0 | 1 | 0
Not completed — Fullfillment of exclusion criteria | 1 | 0 | 0 | 3 | 1
Not completed — Incorrect enrolment or randomization | 4 | 0 | 0 | 0 | 0
Not completed — Interupted IP for more than 7 days | 0 | 4 | 1 | 3 | 3
Not completed — Severe non compliance to protocol | 1 | 0 | 0 | 1 | 2
Not completed — Participant not willing to continue | 7 | 10 | 11 | 5 | 8
Not completed — Criteria from the CSR | 0 | 0 | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3 | Total
Number analyzed (Participants) | 164 | 151 | 156 | 160 | 318 | 949
Age Continuous [Mean (Standard Deviation); unit: Years] | 9.0 (69.9) | 9.0 (69.8) | 9.4 (69.3) | 9.4 (67.8) | 9.1 (68.3) | 9.18 (69.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 49 | 53 | 103 | 299
  Male | 117 | 104 | 107 | 107 | 215 | 650

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Events
Description: Number of patients with a bleeding event while on study drug. Patients with multiple events are counted once
Time Frame: 36 weeks according to protocol. For patients who discontinued treatment the time frame was <36 weeks. Mean number of weeks was 21 weeks (baseline to end of treatment visit)
Measure: Number; unit: Participants
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 164 | 151 | 156 | 160 | 318
Participants | 18 | 8 | 22 | 17 | 46

2. Primary Outcome: Creatinine
Description: Change in Creatinine values from baseline to week 12 visit for patients while on study drug (week 12 visit-baseline)
Time Frame: 12 weeks according to protocol.(baseline to week 12 visit)
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 141 | 132 | 133 | 134 | 298
umol/L | 5.95 (11.18) | 4.81 (12.74) | 7.56 (14.95) | 9.22 (11.24) | 0.43 (11.79)

3. Primary Outcome: Alanine Aminotransferase (ALAT)
Description: Number of patients while on study drug with ALAT>=3 times upper limit of normal.l
Time Frame: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 156 | 147 | 150 | 152 | 315
Participants | 6 | 1 | 5 | 2 | 5

4. Primary Outcome: Bilirubin
Description: Number of patients while on study drug with Bilirubin>=2 times upper limit of normal
Time Frame: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 156 | 147 | 150 | 152 | 315
Participants | 1 | 0 | 0 | 3 | 2

5. Secondary Outcome: D-Dimer
Description: Change in D-Dimer values from enrolment to week 12 visit for VKA naïve patients while on study drug (week 12 visit-enrolment)
Time Frame: 14 weeks according to protocol.(enrolment to week 12 visit)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 37 | 32 | 35 | 43 | 87
ng/mL | -46.4 [-382 to 170] | -76.9 [-613 to 29] | -45.2 [-1817 to 230] | -68.0 [-1313 to 69] | -50.3 [-3955 to 516]

6. Secondary Outcome: Activated Partial Thromboplastin Time (APTT)
Description: Change in Activated partial thromboplastin time (APTT) from baseline to week 12 visit for VKA naïve patients while on study drug (week 12 visit-baseline)
Time Frame: 12 weeks according to protocol.(baseline to week 12 visit)
Measure: Median (Full Range); unit: sec
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 35 | 30 | 34 | 41 | 0
sec | 8.2 [-1 to 24] | 12.3 [2 to 110] | 17.4 [-79 to 52] | 16.4 [2 to 60] |

7. Secondary Outcome: Ecarin Clotting Time (ECT)
Description: Change in Ecarin clotting time (ECT) from baseline to week 12 visit for patients while on study drug (week 12 visit-baseline)
Time Frame: 12 weeks according to protocol.(baseline to week 12 visit)
Measure: Median (Full Range); unit: sec
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 94 | 85 | 85 | 98 | 0
sec | 33.5 [-1 to 86] | 53.0 [15 to 93] | 64.0 [2 to 134] | 73.5 [-1 to 166] |

8. Secondary Outcome: Plasma Concentration of AZD0837 (Prodrug)
Description: Assessment made on the week 12 visit
Time Frame: 12 weeks after baseline according to protocol
Measure: Median (Full Range); unit: nmol/L
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 101 | 104 | 107 | 112 | 0
nmol/L | 199.8 [10.0 to 2334.0] | 617.5 [10.0 to 5355.0] | 564.5 [10.0 to 14720.0] | 1143.5 [10.0 to 9644.0] |

9. Secondary Outcome: Plasma Concentration of AR-H067637XX (Active Metabolite)
Description: Assessment made on the week 12 visit
Time Frame: 12 weeks after baseline according to protocol
Measure: Median (Full Range); unit: nmol/L
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 101 | 104 | 107 | 112 | 0
nmol/L | 223.8 [10.0 to 503.9] | 373.6 [10.0 to 1074.0] | 454.8 [10.0 to 1490.0] | 600.8 [10.0 to 1523.0] |

10. Secondary Outcome: Oral Clearance (CL/F) of AR-H067637XX (Active Metabolite) for C3435T Genotype TT
Description: Oral clearance of AR-H067637XX in subgroup of patients with genotype TT for gene polymorphism ABCB1 C3435T
Time Frame: 36 weeks according to protocol
Measure: Median (Full Range); unit: L/h
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 34 | 41 | 27 | 35 | 0
L/h | 39.7 [22.9 to 79.7] | 42.4 [13.7 to 699] | 36.3 [21.4 to 62.9] | 35.6 [19.7 to 67.3] |

11. Secondary Outcome: Oral Clearance (CL/F) of AR-H067637XX (Active Metabolite) for C3435T Genotype TC
Description: Oral clearance of AR-H067637XX in subgroup of patients with genotype TC for gene polymorphism ABCB1 C3435T
Time Frame: 36 weeks according to protocol
Measure: Median (Full Range); unit: L/h
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 73 | 64 | 64 | 66 | 0
L/h | 39.2 [19.6 to 130.5] | 39.3 [17.2 to 138.6] | 37.7 [18 to 79.4] | 40 [17.4 to 96.7] |

12. Secondary Outcome: Oral Clearance (CL/F) of AR-H067637XX (Active Metabolite) for C3435T Genotype CC
Description: Oral clearance of AR-H067637XX in subgroup of patients with genotype CC for gene polymorphism ABCB1 C3435T
Time Frame: 36 weeks according to protocol
Measure: Median (Full Range); unit: L/h
Arm/Group | 150 mg od | 300 mg od | 450 mg od | 200 mg bd | VKA INR 2-3
Number analyzed (Participants) | 28 | 21 | 31 | 30 | 0
L/h | 40.9 [23.7 to 66] | 41.1 [21.8 to 62.1] | 43.4 [22.8 to 78] | 39.6 [26.5 to 107.1] |

ADVERSE EVENTS:
Arm/Group | AZD0837 150 mg od | AZD0837 300 mg od | AZD0837 450 mg od | AZD0837 200 mg bd | VKA INR 2-3
Serious Adverse Events (participants affected / at risk) | 12/166 | 20/152 | 31/157 | 27/161 | 50/319
Other Adverse Events (participants affected / at risk) | 46/166 | 62/152 | 46/157 | 59/161 | 67/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0837 150 mg od (N=166) | AZD0837 300 mg od (N=152) | AZD0837 450 mg od (N=157) | AZD0837 200 mg bd (N=161) | VKA INR 2-3 (N=319)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 3 | 1 | 1 | 6
Atrial Fibrillation (Cardiac disorders) | 0 | 2 | 4 | 0 | 4
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Angina Unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0 | 1 | 1
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Cardiac Failure Acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1 | 1 | 0 | 1
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 2
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Periodontal Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chest Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Non-Cardiac Chest Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Sudden Death (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Chronic Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Corneal Graft Rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infective Spondylitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Alanine Aminotransferase Increased (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood Glucose Increased (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 2 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope Vasovagal (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Vascular Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Arterial Stenosis Limb (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Axillary Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral Artery Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0837 150 mg od (N=166) | AZD0837 300 mg od (N=152) | AZD0837 450 mg od (N=157) | AZD0837 200 mg bd (N=161) | VKA INR 2-3 (N=319)
DIARRHOEA (Gastrointestinal disorders) | 14 | 23 | 12 | 17 | 15
NAUSEA (Gastrointestinal disorders) | 6 | 8 | 8 | 9 | 15
FLATULENCE (Gastrointestinal disorders) | 10 | 11 | 6 | 10 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 1 | 8 | 2 | 3
NASOPHARYNGITIS (Infections and infestations) | 10 | 10 | 5 | 10 | 20
DIZZINESS (Nervous system disorders) | 4 | 9 | 7 | 11 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less